CLINICAL TRIAL: NCT01592019
Title: Use of Dermal Microdialysis to Evaluate the Effect of Skin Properties and Application Site on the Topical Bioequivalence of Diclofenac: The Main Study
Brief Title: Clinical Study to Evaluate the Role of Microdialysis for the Comparison of Topical Products
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10-223-00277-01
Record Dates: First submitted 2012-04-30; First posted 2012-05-04 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-11

CONDITIONS: Bioequivalence

ARMS (4):
- Reference, Patch location thigh, batch 1 (Experimental): Reference, Patch location thigh, batch 1: A single dose of the patch will be applied. In addition, the Microdialysis probe consisting of three probes will be inserted to test for the amount of the drug diclofenace. This will determine whether the site of application affects the availability of the drug.
  Interventions: Drug: Reference, Patch location thigh, batch 1
- Test, Patch location thigh, batch 2 (Experimental): Test, Patch location thigh, batch 2: A single dose of the patch will be applied. In addition, the Microdialysis probe consisting of three probes will be inserted to test for the amount of the drug diclofenace. This will determine whether the site of application affects the availability of the drug.
  Interventions: Device: Test, Patch location thigh, batch 2
- Reference, Patch location abdomen, batch 1 (Experimental): Reference, Patch location abdomen, batch 1: A single dose of the patch will be applied. In addition, the Microdialysis probe consisting of three probes will be inserted to test for the amount of the drug diclofenace. This will determine whether the site of application affects the availability of the drug.
  Interventions: Drug: Reference, Patch location abdomen, batch 1
- Test, Patch location abdomen, batch 2 (Experimental): Test, Patch location abdomen, batch 2: A single dose of the patch will be applied. In addition, the Microdialysis probe consisting of three probes will be inserted to test for the amount of the drug diclofenace. This will determine whether the site of application affects the availability of the drug.
  Interventions: Device: Test, Patch location abdomen, batch 2

INTERVENTIONS:
Drug: Reference, Patch location thigh, batch 1 — Reference, Patch location thigh, batch 1
  Other Names: Flector patch
  Arms: Reference, Patch location thigh, batch 1
Device: Test, Patch location thigh, batch 2 — Test, Patch location thigh, batch 2. Three probes will be inserted at each visit.
  Other Names: Microdialysis probe
  Arms: Test, Patch location thigh, batch 2
Drug: Reference, Patch location abdomen, batch 1 — Reference, Patch location abdomen, batch 1
  Other Names: Flector Patch
  Arms: Reference, Patch location abdomen, batch 1
Device: Test, Patch location abdomen, batch 2 — Test, Patch location abdomen, batch 2. Three probes will be inserted at each visit.
  Other Names: Microdialysis probe
  Arms: Test, Patch location abdomen, batch 2

SUMMARY:
The investigators hypothesize that a technique called microdialysis can be used to measure the amount of the drug diclofenac which penetrates (enters) the fatty tissue under the skin. Microdialysis uses a small device called a 'probe' to determine the amount of drug which enters a body tissue. The small device is placed directly in the fatty tissue and samples are taken at specific times. The investigators will determine whether site of application affects the availability of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 55 years of age.
* Body mass index of 18.5 and 32 kg/m2, inclusive.
* Non-smoker (not smoked for 12 months prior to screening).
* Healthy on the basis of physical examination, medical history, and vital signs.
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel (including liver enzymes, other specific tests) and hematology are outside the normal reference ranges, the subject may be included only if the study physician judges the abnormalities or deviations from normal to be not clinically significant.
* Female subjects must be postmenopausal (for at least 6 months), surgically sterile, or abstinent; or, if of childbearing potential and sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch) before entry and throughout the study. Also, subjects must have a negative serum human chorionic gonadotropin pregnancy test at the initial screening.
* Agree not to consume any alcohol 72 hours prior to application of the study patch and until discharge from the unit.
* Agree not to use diclofenac-containing medications while enrolled in the study.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Subjects should be willing to shower using the same soap/cleansers between the screening visit and the end of the study, namely the Oil of Olay Moisturizing Bar Soaps with Shea Butter.
* Subjects should be willing avoid the use of body oils, creams, lotions, or powders to the test areas for a period of 48 hours before the application of patches.

Exclusion Criteria:

* Clinically significant abnormal values for hematology or chemistry at screening.
* History of current significant medical illness including (but not limited to) cardiovascular thrombotic events, myocardial infarction, stroke or other cardiac disease, hypertension, peptic ulcer disease or gastrointestinal bleeding, skin disorders, hematological disease, bronchospastic respiratory disease, asthma, diabetes mellitus, renal or hepatic insufficiency, or any other illness that the investigator considers should exclude the subject.
* History of atopic eczema, dry skin or ichthyosis.
* Excessive hair at the site of application that could possibly affect drug absorption; scar tissue, open tissue(s), tattoo or coloration that would interfere with the test sites, their assessments, and their reaction to drug, or that may compromised the safety of the subjects.
* Known allergies or hypersensitivity to Flector® Patch or diclofenac-containing products.
* Clinically significant abnormal physical examination and/or vital signs (e.g. systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg, heart rate >100 bpm and <45 bpm).
* Received an investigational drug (including vaccines) within 60 days prior to study drug administration or are currently enrolled in an investigational study.
* Pregnant or breast-feeding.
* Recent history of surgery; within the past 3 months prior to screening.
* Clinically significant acute illness within 7 days prior to study drug administration.
* Donation of 1 or more units (approximately 450 mL) of blood or acute loss of an equivalent amount of blood within 60 days prior to study drug administration.
* Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.
* Over-the-counter or prescription use of other non-steroidal anti-inflammatory drug products.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Blood and tissue diclofenac concentrations | 24 hours per visit
  Blood and tissue concentrations (nanograms/milliliter) of the drug diclofenac will be measured and compared between different batches of the product Flector. In addition, the two batches will be compared at different application sites, namely the abdomen and thigh. Tissue concentrations will be measured using microdialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Derendorf, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States